CLINICAL TRIAL: NCT02883985
Title: Hypo-Fractionated Conformal Radiation Therapy to the Tumor Bed After Segmental Mastectomy
Brief Title: Safety Study of the Hypo-fractionated (Large Doses) Radiation Therapy in Post-menopausal Women With Breast Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9096
Record Dates: First submitted 2016-08-09; First posted 2016-08-30 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation Therapy: 6 Gy/ fraction (Experimental): All patients will be treated with 6 Gy /fraction delivered in 5 fractions over a 2 week period for a total dose of 30 Gy.
  Interventions: Radiation: 6 Gy/ fraction

INTERVENTIONS:
Radiation: 6 Gy/ fraction — All patients will be treated with 6 Gy (measure of radiation dose) /fraction (each radiation session) delivered in 5 fractions over a 2 week period for a total dose of 30 Gy.
  In addition to routine care, patients may receive antihormonal drugs as part of your base line treatment.

SUMMARY:
The purpose of this study is to determine whether high dose of radiation therapy (RT) are effective over standard 6-week radiation treatment in patients with breast cancer

DETAILED DESCRIPTION:
Hypo-fractionation (several large fractions as the only radiation treatment) for breast cancer irradiation was common in the forties and 50s and, while very successful in achieving tumor control, was found to leave significantly inferior cosmetic results due to severe fibrosis and telangiectasia compared to those obtained with multiple fraction regimens (38-40). These complications were due to the use of very large fields, with the inclusion of a large proportion of uninvolved skin and tissue surrounding the tumor.

Based on these assumptions, a few large fractions can be safely delivered to breast cancers provided that 1) the target volume is sufficiently small and 2) the radiation technique assures maximum sparing of the surrounding normal tissue. Conformal RT to the tumor bed of T1 breast cancers satisfies both requirements.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (at least 2 years without menstrual period):

hysterectomized patients need follicle-stimulating hormone (FSH) confirmation of post-menopausal status.

* Original tumor non-palpable (mammographically detected).
* Small primary tumor (pT1) breast cancer, excised with negative margins (defined as at least a 5 mm margin).
* N0 or sentinel node negative or N0 clinically if the tumor is <1 cm in size.
* Patient offered six weeks of post-segmental mastectomy conventional radiation therapy and declined.
* Prescribed antihormonal therapy as part of their management.

Exclusion Criteria:

* Previous radiation therapy to the ipsilateral breast.
* Presence of a proportion of ductal carcinoma in situ (DCIS) in the pathology specimen which is compatible with extensive intraductal component (EIC).
* Women incapable of providing their own consent. Mental status will be assessed by the Principal Investigator using the Radiation Therapy Oncology Group (RTOG) Mini-Mental Status Examination.
* Women with a diagnosis of multifocal breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-05 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 5 years

SECONDARY OUTCOMES:
TGF-beta 1 determinations | From baseline to up to 4 weeks
  Blood specimens will be collected by venipuncture, before starting treatment, immediately after the last treatment fraction
Ultrasound for target localization | up to 4 weeks
  Ultrasound is ideal for imaging soft tissues unobstructed by bone and has been used successfully in conjunction with the treatment of prostate cancer to verify compliance between the daily location of the prostate and the planned location with respect to the treatment linear accelerator. By using ultrasound to image the post-operative tumor bed of the breast in "real-time", the operator may automatically align the tumor bed with treatment machine on each day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Perez, M.D., Principal Investigator — NYU Perlmutter Cancer Center
Locations (1):
- NYU Perlmutter Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Formenti SC, Hsu H, Fenton-Kerimian M, Roses D, Guth A, Jozsef G, Goldberg JD, Dewyngaert JK. Prone accelerated partial breast irradiation after breast-conserving surgery: five-year results of 100 patients. Int J Radiat Oncol Biol Phys. 2012 Nov 1;84(3):606-11. doi: 10.1016/j.ijrobp.2012.01.039. Epub 2012 Apr 9. PMID 22494589
- See also: Prone accelerated partial breast irradiation after breast-conserving surgery: five-year results of 100 patients — http://www.ncbi.nlm.nih.gov/pubmed/?term=Prone+accelerated+partial+breast+irradiation+after+breast-conserving+surgery%3A+Five+year+results+of+100+patients